CLINICAL TRIAL: NCT02962284
Title: An Open-Label, Single-Arm, Multiple Center Extension Study to Evaluate One Year of Treatment of Patients With Metastatic Castration-Resistant Prostate Cancer With YONSA™ 500 mg (4 x 125 mg qd) With Methylprednisolone (4 mg Bid)
Brief Title: One-year, Open Extension to Evaluate the Treatment of Patients With Castration-Resistant Prostate Cancer With YONSA™
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHL-AA-202
Record Dates: First submitted 2016-10-31; First posted 2016-11-11 (Estimated); Results first posted 2019-07-22 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Abiraterone Acetate; Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YONSA with Methylprednisolone (Experimental): Aberaterone Acetate 500 mg (4 x 125 mg qd) with Methylprednisolone (4 mg bid)
  Interventions: Drug: abiraterone acetate with Methylprednisolone

INTERVENTIONS:
Drug: abiraterone acetate with Methylprednisolone — YONSA 500 mg (4 x 125 mg qd) with Methylprednisolone (4 mg bid)
  Other Names: YONSA

SUMMARY:
This is an open-label, single-arm, multi-center extension study to evaluate safety in patients with mCRPC of YONSA 500 mg (4 x 125 mg qd) with methylprednisolone (4 mg bid). Patients will have successfully completed an 84-day treatment with abiraterone acetate in a previous trial. Results from the final visit of the previous study will be used to determine patient's eligibility for this study. Patients in this study will be eligible to receive open-label YONSA with methylprednisolone for up to 12 months. Pharmacodynamic parameters of serum testosterone and PSA levels will be monitored. Disease progression will be assessed by PCWG2 criteria.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of 84 days of treatment with YONSA in Churchill Pharmaceuticals clinical trial, CHL-AA-201
* Last dose of YONSA or Zytiga within 45 days prior to treatment in this study
* Written informed consent obtained prior to any study-related procedure being performed
* Has in the investigator's opinion, the potential to gain clinical benefit with YONSA treatment
* Ongoing therapy with a GnRH agonist or antagonist AND serum testosterone level <50 ng/dL at screening
* Life expectancy of at least 9 months at screening
* Subject is willing and able to comply with all protocol requirements assessments
* Agrees to protocol-defined use of effective contraception.

Exclusion Criteria:

* Serious concurrent illness, including psychiatric illness, that would interfere with study participation
* Inability to swallow tablets whole
* Known hypersensitivity to YONSA, methylprednisolone, or any excipients in study medications
* Moderate to severe hepatic impairment (Child-Pugh Classes B and C)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Nemeth, Ph.D., Study Director — Churchill Pharmaceuticals LLC

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 20 subjects were enrolled in the study. Of these, 9 subjects were previously treated with YONSA and 11 subjects were previously treated with Zytiga in CHL-AA-201. Twelve (60.0%) subjects completed the study
Groups:
- Preceding Treatment - Yonsa: 84-days treatment: Yonsa 500 mg orally once daily with methylprednisolon
- Preceding Treatment - Zytiga: Yonsa 500 mg orally once daily with methylprednisolon
Period: Overall Study
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Started | 9 | 11
Completed | 4 | 8
Not Completed | 5 | 3
Not completed — Death | 2 | 0
Not completed — Progressive disease | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Preceding Treatment - Yonsa: 84-days treatment
- Preceding Treatment - Zytiga: 84 day treatment
- Total: Total of all reporting groups
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Customized [Count of Participants; unit: Participants]
  <75 years | 4 | 5 | 9
  ≥75 years | 5 | 6 | 11
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 7 | 11 | 18
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events
Description: Adverse events
Time Frame: one year
Population: subjects who were enrolled and who received at least 1 dose of study drug of Yonsa
Measure: Number; unit: Participants
Groups:
- Preceding Treatment - Yonsa; Preceding Treatment - Zytiga: one year treatment
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 9 | 11
Participants | 8 | 9

2. Secondary Outcome: Proportion of Subjects With Disease Progression
Description: Number of participants who had disease progression
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 9 | 11
Participants | 1 | 3
Statistical Analysis 1: Comparison: Preceding Treatment - Yonsa vs Preceding Treatment - Zytiga; Test type: Superiority; p > 0.1, ANCOVA

3. Secondary Outcome: Testosterone Levels
Description: Change in serum testosterone levels from baseline
Time Frame: Baseline and 360 days
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 3 | 6
ng/dL | -6.24 (2.02) | -5.87 (3.64)

4. Secondary Outcome: Prostate Specific Antigen Levels
Description: Change in serum testosterone levels after one year of treatment against baseline
Time Frame: One year
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 5 | 9
ng/dL | -60.12 (115.63) | -112.76 (239.85)

5. Secondary Outcome: Testosterone Complete Suppression
Description: Proportion of subjects with complete suppression of testosterone levels
Time Frame: 360 days
Measure: Number; unit: percentage of subjects
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 5 | 8
percentage of subjects | 100 | 87.5

6. Secondary Outcome: Percentage of Subjects With Prostate Specific Antigen - 50 Response
Description: A decrease of ≥50% reduction from baseline of the study CHL-AA-201
Time Frame: 360 days
Measure: Number; unit: percentage of number of subjects
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
Number analyzed (Participants) | 5 | 9
percentage of number of subjects | 60.0 | 55.6

ADVERSE EVENTS:
Time Frame: One year
Arm/Group | Preceding Treatment - Yonsa | Preceding Treatment - Zytiga
All-Cause Mortality (participants affected / at risk) | 2/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/11
Other Adverse Events (participants affected / at risk) | 8/9 | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preceding Treatment - Yonsa (N=9) | Preceding Treatment - Zytiga (N=11)
Septic shock (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Abasia (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Right leg cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preceding Treatment - Yonsa (N=9) | Preceding Treatment - Zytiga (N=11)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
-Dry mouth (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Abasia (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 1
Mass (General disorders) | 1 | 0
Nodule (General disorders) | 1 | 0
Non-cardiac chest pai (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 1 | 1
Ulcer (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-02): https://cdn.clinicaltrials.gov/large-docs/84/NCT02962284/Prot_SAP_000.pdf